CLINICAL TRIAL: NCT00484666
Title: A Phase II Study of Weekly Docetaxel and Topotecan in Patients With Platinum-Resistant, Recurrent Epithelial Ovarian Cancer
Brief Title: Platinum-Resistant, Recurrent Epithelial Ovarian Cancer
Acronym: TopoTxt
Status: Withdrawn | Type: Observational
Why Stopped: PI withdrew from study protocol participation
Sponsor: Carilion Clinic (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: Topo Txt
Record Dates: First submitted 2007-06-07; First posted 2007-06-11 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Ovarian Cancer
Keywords: recurrent; platinum; resistant; ovarian; primary; peritoneal; cancer
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Primary objective:

To estimate the overall clinical response rate (CR, PR, SD) of weekly docetaxel and weekly topotecan in women with recurrent platinum resistant ovarian or primary peritoneal cancer.

Secondary objectives:

To access the safety and tolerability of this novel combination chemotherapy regimen of weekly docetaxel and weekly topotecan in women with recurrent platinum resistant ovarian or primary peritoneal cancer

To estimate the progression free survival (PFS) and overall survival (OS) for women with recurrent platinum resistant ovarian or primary peritoneal cancer treated with this weekly docetaxel and weekly topotecan.

DETAILED DESCRIPTION:
Each year more than 28,000 women are diagnosed with epithelial ovarian cancer (EOC). Over 70% of these women will present with advanced (stage III, IV) disease. The current treatment for newly diagnosed advanced EOC involves cytoreductive surgery followed by chemotherapy. The standard chemotherapy in the primary setting is a combination of a taxane; either paclitaxel or docetaxel and a platinum agent; either cisplatin or carboplatin. Although high initial responses are seen with these primary therapies, most will recur. Salvage chemotherapy thus becomes the mainstay of treatment for many patients with this disease. The goals of salvage therapy are to maximize tumor response while maintaining quality of life with minimal toxicity. As a consequence, there are a number of agents that have been studied in this recurrent setting with significant antitumor activity. Two such novel agents, topotecan and docetaxel are the basis of this phase I, II study.

Patients can be grouped into prognostic categories based on their responses to primary therapy. Those with persistent disease or recurrence within 6 months of treatment are deemed platinum resistant and those achieving a greater than 6 month progression free interval are deemed platinum sensitive. This distinction is important because those that are platinum sensitive have an improved overall survival and higher response rates to salvage chemotherapy. The magnitude of this response increases with an increasing progression free interval. The response of these patients to reintroducing either platinum or paclitaxel has been established. Thigpen et. al. showed a 44% overall response rate(ORR) to paclitaxel infused over 24 hours in 16 patients with a platinum free interval of greater than or equal to 6 months. Kavanagh et. al. demonstrated a 21% partial response rate (PR) to the reintroduction of carboplatin after taxane treatment in 26 patients with a 12-month platinum-free intraval following platinum-refractory ovarian cancer.

Topotecan has been shown to have similar activity as paclitaxel as a second line therapy with non-cross resistance. Topotecan is usually administered in a daily infusion over 30 minutes in doses of 1.5 mg/m2/d x 5 consecutive days every 21 days. In an effort to decrease toxicity and maintain response rates, weekly schedules of topotecan have been explored. Homesley et. al. conducted a phase I trial with single agent weekly topotecan evaluating dosages from 1.5 to 6 mg/m2/wk. The recommended phase II dosage for weekly topotecan was determined to be 4 mg/m2/wk. Dose limiting toxicities consisted of 70 non-hematologic events in 32 of 35 evaluable patients, primarily consisting of grade 1 or 2 chronic fatigue (16%) and gastrointestinal (nausea and vomiting [23%]) with the majority (80%) being grade 1 in severity. Dose limiting myelotoxicity and thrombocytopenia were not an issue at the weekly dosages evaluated in this trial. Morris and colleagues at Wayne State University are currently studying weekly topotecan in platinum sensitive patients and have reported a 40% partial response rate with 35% having stable disease. Myelotoxicity was infrequent and included grade 3 or 4 neutropenia in 1.1% and grade 3 anemia in 1.8%. Nonhematologic toxicity included grade 3 fatigue in 17% of patients.

Abu-Rustum et. al. conducted a phase I trial of weekly paclitaxel (60 -100 mg/m2 over 1-hour) in platinum resistant patients (n = 18 patients, recommended phase II dose 80 mg/mg/wk). Dose limiting toxicity was defined as two or more patients with treatment delay or grade 3 toxicity at the same dose level. Treatment was delayed in 2 of 3 patients at the 100 mg/m2 dose level due to ANC < 1500. In addition they reviewed Memorial Sloan Kettering's previous data with weekly paclitaxel (60 to 100 mg/m2/wk) in platinum resistant patients and found an overall response rate (either documented tumor shrinkage or decrease in serum CA-125 levels) of 28% (ORR in 13 of 45 patients). In a follow up phase II trial, Markman et. al. reported a 25% objective response rate in 13 of 51 platinum resistant patients (4 by decreasing CA-125 and 9 by 50% reduction in tumor volume). Only 1% (13 of 887 dosages) required a dose modification due to toxicity with weekly paclitaxel at 80 mg/m2/wk. Weekly paclitaxel is an active second-line regimen and is generally well tolerated.

In advanced, platinum-refractory ovarian cancer, docetaxel administered every 3 weeks has demonstrated substantial single-agent efficacy with response rates ranging from 24% to 40% and an overall survival of 8 to 10.4 months. Neutropenia was the predominant Grade 3 /4 toxicity, followed by fluid retention, hypersensitivity reactions and diarrhea.

The combination of docetaxel and carboplatin has been studied as first-line therapy for the treatment of epithelial ovarian cancer. A phase II study by Markman et.al. utilized docetaxel 60 mg/m2 plus carboplatin AUC 6 every 3 weeks demonstrated an overall response rate of 81%. The most common hematologic toxicity was Grade 4 neutropenia (64%), while neutropenic fever was observed in only 6% of those patients. The most common non-hematologic toxicity was a mild hypersensitivity reaction (34%) that did not prevent patients from completing their planned therapy.

Preliminary results have recently been reported from a randomized phase III trial comparing docetaxel (75 mg/m2/1 hr infusion) to paclitaxel (175 mg/m2/3 hr infusion) in combination with carboplatin (AUC 5 as calculated by 51Cr-EDTA secretion) every 3 weeks as first-line chemotherapy following surgery for Stage Ic-IV ovarian cancer. Both combinations demonstrated very high overall response rates of 65% and 62%, respectively, and an estimated 1 year disease free survival is approximately 60% for both treatment groups. With regard to toxicity, the occurrence of Grade 2-4 sensory neurotoxicity was significantly increased in patients receiving paclitaxel (30%) compared to docetaxel (11%; p<.001) and accounted for the majority of toxicity related treatment withdrawal in the paclitaxel group. The most common severe side effect was myelosuppression with Grade 3 or 4 neutropenia occurring in 84% of patients treated with paclitaxel and 94% of patients treated with docetaxel (p<.001). Febrile neutropenia was noted in 10% of patients treated with docetaxel, compared to 2% of patients treated with paclitaxel (p<.001). However, there was no difference in septic mortality between the two treatment arms.

In order to decrease the incidence of hematological toxicity associated with docetaxel administered every three weeks, clinicians have explored the use of docetaxel on a weekly schedule. There have been numerous published reports examining the role of weekly docetaxel (single agent and in combination chemotherapy regimens) in wide range of solid tumors including breast, NSCLC, prostate and ovarian. Weekly administration of docetaxel resulted in substantial clinical activity, was well tolerated and resulted in a decreased incidence of hematologic toxicity (grade 3/4 neutropenia and leukopenia each reported in ≤16% of patients; grade 3/4 anemia and thrombocytopenia in ≤13% and ≤3% of patients, respectively. Acute toxicities were uncommon, as was peripheral neuropathy. Prolonged treatment with weekly docetaxel results in chronic toxicities, including asthenia (fatigue), edema, tearing (excessive lacrimation or epiphora), and nail changes. Chronic toxicities have been most prominent when docetaxel has been administered on a continuous weekly basis, i.e., without a break. Toxicities appeared to be delayed in onset or avoided by providing treatment breaks. The current strategy is treating weekly 2 out of 3 weeks on an every 21-day cycle or weekly 3 out of 4 weeks on an every 28-day cycle. The reduced incidence of myelosuppression may enhance the feasibility and tolerability of weekly docetaxel-containing combination regimens.

Burris and colleagues have enrolled 36 patients in a phase I study of weekly docetaxel (20, 25, 30 mg/m2/wk) and weekly topotecan (2.0, 3.0, 3.5 to 4 mg/m2/wk) for solid tumors. The combination of weekly docetaxel 30 mg/m2/wk plus topotecan 3 mg/m2/wk on days 1, 8 and 15 every 28 days resulted in no dose-limiting toxicities and no dose reductions or treatment omissions were warranted during cycle 1 of therapy. Non-hematologic toxicities consisted of grade 1 and 2 nausea, vomiting, fatigue and weakness. Dose-limiting toxicity was documented for weekly docetaxel 30 mg/m2/wk plus topotecan 4 mg/m2/wk with two patients experiencing day 15 dose omissions (one patients with platelets 53 K and ANC 500 and one patient with platelets 27 K who was previously treated with oxaliplatin. Eleven patients have been treated to date with weekly docetaxel 30 mg/m2/wk plus topotecan 3.5 mg/m2/wk. Two patients were non-evaluable, one due to rapidly progressive disease and one due to noncompliance. Of the nine evaluable patients, five patients experienced dose-limiting toxicities as follows, (1) cycle 1 day 15 (C1D15) held due to platelets 33K in a heavily pretreated patient, including previous oxaliplatin, (2) C1D15 dose decreased due to grade 3 diarrhea, (3) C1D8 held due to grade 3-4 nausea and vomiting (may have been disease related), (4) C1D15 held due to platelets 49 K (74 yo, heavily pretreated including previous XRT), (5) C1D15 held due to platelets 43K and declining creatinine clearance of 43 ml/min (3 prior regimens, including XRT, PS 2 and history of thrombocytopenia). One additional patient is planned to complete this dose level, to provide 10 evaluable patients. Of the 36 patients receiving 76 cycles of therapy, myelosuppression was brief and reversible with no febrile neutropenia. Per verbal communication from Dr. Burris, the recommended phase II dose will be docetaxel 30 mg/m2/wk plus topotecan 3.5 mg/m2/wk on days 1, 8 and 15 every 28 days for minimally pretreated patients.

Given the results of these data and the goal to increase response rates in platinum resistant recurrent EOC patients it would seem prudent to evaluate the safety and efficacy of weekly docetaxel 30 mg/m2/wk plus weekly topotecan 3.5 mg/m2/wk via a phase II trial. Results of this trial will be important by expanding our current knowledge base utilizing weekly scheduling of chemotherapeutic agents in regard to toxicities and response rates in platinum resistant EOC.

ELIGIBILITY:
Inclusion Criteria:

* All patients will have had histologically documented ovarian epithelial, fallopian tube or peritoneal cancer.
* Patients must have received one prior platinum- and paclitaxel based regimen
* Patients must be platinum-resistant defined as recurrence or progression of disease <6 months since previous treatment with a platinum based treatment regimen.
* Patients must not have received radiotherapy.
* Patients with the following histologic epithelial cell types are eligible:

  * Serous Adenocarcinoma
  * Endometrioid Adenocarcinoma
  * Mucinous Adenocarcinoma
  * Undifferentiated carcinoma
  * Clear cell Adenocarcinoma
  * Mixed epithelial carcinoma
  * Transitional cell
  * Malignant Brenner's tumor
  * Adenocarcinoma NOS
* Patients may have measurable or evaluable disease whereas evaluable disease is defined as new onset pleural effusion, ascites or a rise in CA-125 level >2x institutions upper limit of normal x 2 now sooner than one week apart.
* Patients could not have more than two previous chemotherapeutic regimens for their advanced ovarian cancer.
* Patients must be at least 18 years of age
* Patients must have a serum creatinine < 1.5 mg/dl
* Patients must have adequate hematologic reserve (ANC > 1500/mm3, hemoglobin ≥ 9.0 gm/dL and platelets > 100,000/mm3)
* Patients must have adequate hepatocellular function:

  * Total Bilirubin < institutional upper limits of normal (ULN), AST or ALT and Alkaline Phosphatase must be within the range allowing for eligibility
* Patients must have GOG performance status of 0, 1 or 2.
* Patients must a have signed, approved informed consent form on file.

Exclusion Criteria:

* Patients with borderline ovarian cancer.
* Patients with GOG performance status 3 or 4.
* Patients who have received prior topotecan and/or docetaxel.
* Patients who have a history of psychiatric illness or other concurrent severe and/or uncontrolled co-morbid medical condition that would preclude study completion (i.e., uncontrolled infection, hypertension, ischemic heart disease, myocardial infarction within 6 months, congestive heart failure).
* Patients with other invasive malignancies, with the exception of non-melanoma skin cancer or any evidence of the other cancer(s) present within the last 5 years or whose previous cancer treatment contraindicates this protocol therapy.
* Patients with a history of severe acute hypersensitivity reaction to medications formulated with polysorbate 80.
* Patients with baseline peripheral neuropathy ≥ Grade 2.
* No use of investigational drugs or alternative medicine anticancer therapy within the last 4 weeks of 1st dose of study drug.
* Pregnant or lactating women with reproductive potential. (All patients enrolled in this study will be postmenopausal or have undergone surgery that includes hysterectomy and oophorectomy that would render them unable to conceive children.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological sex based
Study Population: Females over 18 years of age
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-05 (Actual); Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To estimate the overall clinical response rate (CR, PR, SD) of weekly docetaxel and weekly topotecan in women with recurrent platinum resistant ovarian or primary peritoneal cancer. | 12 Months

SECONDARY OUTCOMES:
To access the safety and tolerability of this novel combination chemotherapy regimen of weekly docetaxel and weekly topotecan in women with recurrent platinum resistant ovarian or primary peritoneal cancer | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Dennis R Scribner, JR, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion GYN Oncology Associates, Roanoke, Virginia, United States

REFERENCES:
- [Background] Neijt JP, Engelholm SA, Tuxen MK, Sorensen PG, Hansen M, Sessa C, de Swart CA, Hirsch FR, Lund B, van Houwelingen HC. Exploratory phase III study of paclitaxel and cisplatin versus paclitaxel and carboplatin in advanced ovarian cancer. J Clin Oncol. 2000 Sep;18(17):3084-92. doi: 10.1200/JCO.2000.18.17.3084. PMID 10963636
- [Background] Papadimitriou CA, Moulopoulos LA, Vlahos G, Voulgaris Z, Kiosses E, Georgoulias N, Gika D, Diakomanolis E, Michalas S, Dimopoulos MA. Paclitaxel, cisplatin, and epirubicin first-line chemotherapy in stage III and IV ovarian carcinoma: long-term results of a phase II study. Cancer. 2000 Oct 1;89(7):1547-54. doi: 10.1002/1097-0142(20001001)89:73.0.co;2-p. PMID 11013370
- [Background] Ozols RF, Bundy BN, Fowler J, Clarke-Pearson D, Mannel R, Hartenbach EM, Baergen R. Randomized phase III study of cisplatin/paclitaxel versus carboplatin/paclitaxel in optimal stage III epithelial ovarian cancer: A GOG trial. Proc Am Soc Clinic Onc 1999;18:356a.
- [Background] Berek JS, Bertelsen K, du Bois A, Brady MF, Carmichael J, Eisenhauer EA, Gore M, Grenman S, Hamilton TC, Hansen SW, Harper PG, Horvath G, Kaye SB, Luck HJ, Lund B, McGuire WP, Neijt JP, Ozols RF, Parmar MK, Piccart-Gebhart MJ, van Rijswijk R, Rosenberg P, Rustin GJ, Sessa C, Willemse PH, et al. Advanced epithelial ovarian cancer: 1998 consensus statements. Ann Oncol. 1999;10 Suppl 1:87-92. doi: 10.1023/a:1008323922057. PMID 10219460
- [Background] Markman M, Rothman R, Hakes T, Reichman B, Hoskins W, Rubin S, Jones W, Almadrones L, Lewis JL Jr. Second-line platinum therapy in patients with ovarian cancer previously treated with cisplatin. J Clin Oncol. 1991 Mar;9(3):389-93. doi: 10.1200/JCO.1991.9.3.389. PMID 1999708
- [Background] Thigpen JT, Blessing JA, Ball H, Hummel SJ, Barrett RJ. Phase II trial of paclitaxel in patients with progressive ovarian carcinoma after platinum-based chemotherapy: a Gynecologic Oncology Group study. J Clin Oncol. 1994 Sep;12(9):1748-53. doi: 10.1200/JCO.1994.12.9.1748. PMID 7916038
- [Background] Kavanagh J, Tresukosol D, Edwards C, Freedman R, Gonzalez de Leon C, Fishman A, Mante R, Hord M, Kudelka A. Carboplatin reinduction after taxane in patients with platinum-refractory epithelial ovarian cancer. J Clin Oncol. 1995 Jul;13(7):1584-8. doi: 10.1200/JCO.1995.13.7.1584. PMID 7602347
- [Background] Gore M, ten Bokkel Huinink W, Carmichael J, Gordon A, Davidson N, Coleman R, Spaczynski M, Heron JF, Bolis G, Malmstrom H, Malfetano J, Scarabelli C, Vennin P, Ross G, Fields SZ. Clinical evidence for topotecan-paclitaxel non--cross-resistance in ovarian cancer. J Clin Oncol. 2001 Apr 1;19(7):1893-900. doi: 10.1200/JCO.2001.19.7.1893. PMID 11283120
- [Background] Homesley HD, Hall DJ, Martin DA, Lewandowski GS, Vaccarello L, Nahhas WA, Suggs CL, Penley RG. A dose-escalating study of weekly bolus topotecan in previously treated ovarian cancer patients. Gynecol Oncol. 2001 Nov;83(2):394-9. doi: 10.1006/gyno.2001.6435. PMID 11606103
- [Background] Morris RT, Munkarah A, Field J, Baker VV, Drake R, Malone J. Phase II trial of weekly topotecan in patients with potentially platinum sensitive relapsed ovarian and peritoneal cancer. Proc ASCO, 2002; 2512A.
- [Background] Abu-Rustum NR, Aghajanian C, Barakat RR, Fennelly D, Shapiro F, Spriggs D. Salvage weekly paclitaxel in recurrent ovarian cancer. Semin Oncol. 1997 Oct;24(5 Suppl 15):S15-62-S15-67. PMID 9346225
- [Background] Markman M, Hall J, Spitz D, Weiner S, Carson L, Van Le L, Baker M. Phase II trial of weekly single-agent paclitaxel in platinum/paclitaxel-refractory ovarian cancer. J Clin Oncol. 2002 May 1;20(9):2365-9. doi: 10.1200/JCO.2002.09.130. PMID 11981009
- [Background] Aapro MS, Pujade-Lauriane E, et al. EORTC Clinical Screening Group: Phase II study of Taxotere in ovarian cancer. Annals of Oncology 5(5):202, abstract 508, 1994.
- [Background] Francis P, Schneider J, Hann L, Balmaceda C, Barakat R, Phillips M, Hakes T. Phase II trial of docetaxel in patients with platinum-refractory advanced ovarian cancer. J Clin Oncol. 1994 Nov;12(11):2301-8. doi: 10.1200/JCO.1994.12.11.2301. PMID 7964944
- [Background] Kavanagh JJ, Kudelka AP, de Leon CG, Tresukosol D, Hord M, Finnegan MB, Kim EE, Varma D, Forman A, Cohen P, Edwards CL, Freedman RS, Verschraegen CF. Phase II study of docetaxel in patients with epithelial ovarian carcinoma refractory to platinum. Clin Cancer Res. 1996 May;2(5):837-42. PMID 9816238
- [Background] Piccart MJ, Gore M, Ten Bokkel Huinink W, Van Oosterom A, Verweij J, Wanders J, Franklin H, Bayssas M, Kaye S. Docetaxel: an active new drug for treatment of advanced epithelial ovarian cancer. J Natl Cancer Inst. 1995 May 3;87(9):676-81. doi: 10.1093/jnci/87.9.676. PMID 7752272
- [Background] Markman M, Kennedy A, Webster K, Peterson G, Kulp B, Belinson J. Combination chemotherapy with carboplatin and docetaxel in the treatment of cancers of the ovary and fallopian tube and primary carcinoma of the peritoneum. J Clin Oncol. 2001 Apr 1;19(7):1901-5. doi: 10.1200/JCO.2001.19.7.1901. PMID 11283121
- [Background] Vasey PA, Atkinson R, Coleman R, Crawford M, Cruickshank M, Eggleton P, Fleming D, Graham J, Parkin D, Paul J, Reed NS, Kaye SB. Docetaxel-carboplatin as first line chemotherapy for epithelial ovarian cancer. Br J Cancer. 2001 Jan;84(2):170-8. doi: 10.1054/bjoc.2000.1572. PMID 11161372
- [Background] Vasey PA et. al. Proc Am Soc Clin Onc 2001;20:Abst.1370.
- [Background] Kuzur ME, Jones S, Willcutt N, et al. The Sarah Cannon Cancer Center/Tennessee Oncology, Nashville, TN; Glaxo Smith Kline, Philadelphia, PA: A phase I trial of weekly topotecan and docetaxel. Proc Am Soc Clin Onc 2003;22:Abst.
- [Background] Hainsworth JD, Burris HA 3rd, Erland JB, Thomas M, Greco FA. Phase I trial of docetaxel administered by weekly infusion in patients with advanced refractory cancer. J Clin Oncol. 1998 Jun;16(6):2164-8. doi: 10.1200/JCO.1998.16.6.2164. PMID 9626217
- [Background] Burstein HJ, Manola J, Younger J, Parker LM, Bunnell CA, Scheib R, Matulonis UA, Garber JE, Clarke KD, Shulman LN, Winer EP. Docetaxel administered on a weekly basis for metastatic breast cancer. J Clin Oncol. 2000 Mar;18(6):1212-9. doi: 10.1200/JCO.2000.18.6.1212. PMID 10715290
- [Background] Stemmler J, Mair W, Stauch M, et al. Weekly docetaxel with or without corticosteroid premedication as first or second-line treatment in patients (pts) with metastatic breast cancer (MBC). Proc Am Soc Clin Oncol. 2002;21:58a. Abstract 231.
- [Background] Hainsworth JD, Burris HA 3rd, Yardley DA, Bradof JE, Grimaldi M, Kalman LA, Sullivan T, Baker M, Erland JB, Greco FA. Weekly docetaxel in the treatment of elderly patients with advanced breast cancer: a Minnie Pearl Cancer Research Network phase II trial. J Clin Oncol. 2001 Aug 1;19(15):3500-5. doi: 10.1200/JCO.2001.19.15.3500. PMID 11481356
- [Background] Climent MA, Tabernero J, Albanell J, et al. Preliminary results of a phase II randomized trial of docetaxel (taxotere) as a single agent chemotherapy (CT) administered weekly or 3-weekly in patients (pts) with metastatic breast cancer (MBC). Proc Am Soc Clin Oncol.2002;21:52a. Abstract 205.
- [Background] Hainsworth JD, Burris HA 3rd, Litchy S, Morrissey LH, Barton JH, Bradof JE, Greco FA. Weekly docetaxel in the treatment of elderly patients with advanced nonsmall cell lung carcinoma. A Minnie Pearl Cancer Research Network Phase II Trial. Cancer. 2000 Jul 15;89(2):328-33. doi: 10.1002/1097-0142(20000715)89:23.0.co;2-f. PMID 10918162
- [Background] Lilenbaum RC, Schwartz MA, Seigel L, Belette F, Blaustein A, Wittlin FN, Davila E. Phase II trial of weekly docetaxel in second-line therapy for nonsmall cell lung carcinoma. Cancer. 2001 Oct 15;92(8):2158-63. doi: 10.1002/1097-0142(20011015)92:83.0.co;2-2. PMID 11596033
- [Background] McKay C III, Hainsworth J, Burris H III, et al. Weekly docetaxel/gemcitabine in the treatment of elderly patients (pts) with advanced non-small cell lung cancer (NSCLC): a Minnie Pearl Cancer Research Network phase II trial. Proc Am Soc Clin Oncol. 2001;20:260b. Abstract 2793.
- [Background] Gervais R, Ducoloné AMD, Breton J-L, et al. Multicenter, randomised, phase II trial of docetaxel (Taxotere) 75 mg/m2 q3w versus 40 mg/m2 weekly in patients with pretreated non small cell lung cancer (NSCLC). Proc Am Soc Clin Oncol. 2002;21:310a. Abstract 1238.
- [Background] Schütte W, Nagel S, Lautenschläger C, et al. Randomized phase III study of weekly versus three-weekly docetaxel as second-line chemotherapy for advanced non-small cell lung cancer (NSCLC). Proc Am Soc Clin Oncol. 2002;21:308a. Abstract 1228.
- [Background] Kuzur, ME, Jones S, Willcutt N, et.al. A phase I trial of weekly topotecan and docetaxel. Proc Am Soc Clin Oncol. 2003;22: Abstract 2840.
- [Background] Hycamtin (topotecan) package insert. GlaxoSmithKline. Research Triangle Park, NC. Revised 11/2002.
- [Background] Taxotere (docetaxel) package insert. Aventis Pharmaceuticals, Inc. Bridgewater, NJ. Revised: April/2003.